CLINICAL TRIAL: NCT02927665
Title: A Prospective Multicenter Post Approval Study of the ReShape™ Integrated Dual Balloon System in Obese Subjects
Acronym: ReShapePAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ReShape Post Approval Study
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Obesity
Keywords: Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Subjects: Eligible subjects receiving ReShape Integrated Dual Balloon System treatment in a commercial clinical setting
  Interventions: Device: Reshape Integrated Dual Balloon

INTERVENTIONS:
Device: Reshape Integrated Dual Balloon
  Other Names: Reshape Integrated Dual Balloon System

SUMMARY:
The ReShape Post Approval Study is a prospective multicenter study of the ReShape(TM) Integrated Dual Balloon System in Obese Subjects.

DETAILED DESCRIPTION:
The ReShape Post Approval Study is a post-approval, multicenter, single arm, open label clinical study intended to collect valid scientific evidence regarding the safety and efficacy of the ReShape Dual Balloon as an adjunct to diet and exercise in the treatment of BMI 30-40 subjects with one or more obesity-related comorbid conditions in a commercial clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 22 and older
2. Baseline BMI 30 - 40
3. Failed weight reduction with diet and exercise alone
4. One or more obesity-related comorbid conditions
5. If female of child bearing potential, willing to avoid pregnancy during course of treatment

Exclusion Criteria:

1. Prior gastrointestinal surgery with sequelae, i.e. obstruction, and/or adhesive peritonitis or known abdominal adhesions
2. Prior open or laparoscopic bariatric surgery.
3. Any inflammatory disease of the gastrointestinal tract including esophagitis, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease.
4. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses.
5. A gastric mass.
6. A hiatal hernia > 5 cm or ≤ 5 cm with associated severe or intractable gastro-esophageal reflux symptoms.
7. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the delivery catheter and/or an endoscope.
8. Achalasia or any other severe esophageal motility disorder that may pose a safety risk during the removal of the device
9. Severe coagulopathy
10. Hepatic insufficiency or cirrhosis
11. Serious or uncontrolled psychiatric illness or disorder that could compromise patient understanding of or compliance with follow up visits and removal of the device after 6 months.
12. Alcoholism or drug addiction.
13. Patients unwilling to participate in an established medically-supervised diet and behavior modification program, with routine medical follow-up.
14. Patients receiving daily prescribed treatment with aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants.
15. Patients who are unable or unwilling to take prescribed proton pump inhibitor medication for the duration of the device implant.
16. Patients who are known to have, or suspected to have, an allergic reaction to materials contained in the system.
17. Patients who have ever developed a serotonin syndrome and are currently taking any drug known to affect the levels of serotonin in the body [e.g., selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MAOIs)] should not undergo placement of the device.
18. Patients who are pregnant or breast-feeding.
19. Significant endoscopic abnormalities immediately prior to device insertion.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with a body mass index (BMI) of 30-40 and one or more obesity-related comorbid conditions, who have failed weight reduction with diet and exercise alone
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2016-09; Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Safety of ReShape Dual Balloon Treatment | 24 weeks
  Safety of ReShape Dual Balloon Treatment using a composite endpoint consisting of all device- and/or procedure-related SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shikora, Study Director — ReShape Lifesciences
Locations (14):
- United States (14):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Christiana Institute of Advanced Surgery, Newark, Delaware
  - Barrington Surgeons, Barrington, Illinois
  - The Gastro Clinic, Lafayette, Louisiana
  - Surgical Specialist of Louisiana, Metairie, Louisiana
  - Washington University, St Louis, Missouri
  - North Jersey Laparoscopic Associates, Teaneck, New Jersey
  - New York Bariatric Group, Roslyn Heights, New York
  - JourneyLite Physicians, Cincinnati, Ohio
  - Salem General Surgery, Salem, Ohio
  - Gastrointestinal Associates, P.C., Knoxville, Tennessee
  - MidSouth Bariatrics, Memphis, Tennessee
  - Sage Bariatric Institute, San Antonio, Texas
  - Eviva, Shoreline, Washington

IPD SHARING:
Plan to Share IPD: No